CLINICAL TRIAL: NCT03772717
Title: Non-invasive Vagus Nerve Stimulation (nVNS) in Pediatric Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated due to difficulties with enrollment and poor adherence to the study intervention among participants.
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Sumit Verma, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00098592
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Pediatrics; Vagus nerve stimulation
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Non-invasive vagus nerve stimulation (nVNS) (Experimental): Participants will use the electrical neuromuscular stimulator device, VitalStim 400, which has been used in previous clinical studies for modulation of pain and has received FDA approval. Participants will also continue to take their standard of care medication.
  Interventions: Device: Non-invasive vagus nerve stimulation (nVNS); Other: Standard of care treatment

INTERVENTIONS:
Device: Non-invasive vagus nerve stimulation (nVNS) — The nVNS study intervention will be delivered using a handheld electrical neuromuscular stimulator device (VitalStim 400). Participants will deliver nVNS twice per day for 60 minutes each time at least 5 days per week. The two electrodes for the device will be placed on the subjects left cervical (neck) region. Parents will be trained on where to place electrodes, how to ensure that the electrodes make a good contact with the skin, and how to set the stimulation parameters. The stimulation frequency (number of pulses) and amplitude (amount of current) will be set during the initial baseline session in the clinic at a level that prevents discomfort and does not impact cardiorespiratory parameters. The stimulator will be placed in a comfortable position, such as next to the pillow. The stimulators are battery-powered and allow configuration of the stimulation parameters to the comfort of the patient.
  Other Names: VitalStim 400
Other: Standard of care treatment — Patients will be asked to continue their standard medication regimens which include in most cases will involve 3 weekly infusions of intravenous immunoglobulin (IVIG) (1 gm/kg) and rarely plasma exchange (PLEX).
  Other Names: intravenous immunoglobulin (IVIG); plasma exchange (PLEX)

SUMMARY:
Participants will be requested to deliver non-invasive vagus nerve stimulation (nVNS) two times per day, at least five days per week. Participants will be followed for two years with nVNS as an adjunctive therapy to the standard of care therapy for chronic inflammatory demyelinating polyneuropathy (CIDP).

DETAILED DESCRIPTION:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a chronic immune-mediated disease of the peripheral sensory motor nerves characterized by motor weakness, sensory loss, muscle wasting and loss of motor ability. The majority of CIDP cases are idiopathic with insidious onset, relapsing remitting course, and a prolonged clinical course (over years). CIDP incidence is unknown in pediatric population, however, it is a rare treatable cause of neuromuscular weakness in children. Treatment of CIDP involves chronic use of steroids, intravenous immunoglobulin (IVIG) and, rarely, plasma exchange (PLEX). Despite above mentioned treatments the majority of patients continue to have tremendous disease burden. There is a need for alternative or adjunctive therapies that can decrease chronic inflammation effectively and safely in pediatric CIDP patients.

Vagus nerve stimulation has received significant scientific and clinical attention and has been shown to effectively reduce systemic inflammation. Results from early clinical trials for treatment of Rheumatoid Arthritis (RA) have demonstrated significant lifestyle benefits and reduced symptoms in RA patients. Similar benefits of VNS have been observed in Crohn's disease patients. In these studies, patients are surgically implanted with a stimulator and electrodes directly on the nerve. Preliminary results have demonstrated safety and efficacy in patients that previously were unresponsive to traditional pharmacological therapies. Unfortunately, surgical implantation of a device is difficult and costly.

Recent investigations have significantly increased the understanding of non-invasive vagus nerve stimulation (nVNS). Compared to traditional implanted vagus nerve stimulation devices, nVNS uses electrodes placed on the skin surface to stimulate the vagus nerve. nVNS has shown promise in animal and human models to reduce chronic inflammation in multiple disease states. By delivering electrical pulses at the skin surface above the vagus nerve, neural pathways involved in regulating systemic inflammation are activated. Using a handheld device, patients apply brief durations of stimulation multiple times per day to achieve therapeutic benefit. nVNS is currently FDA approved for clinical use in the treatment of migraines and cluster headaches, with on-going clinical studies on epilepsy and systemic inflammation. Preliminary published results have demonstrated significant therapeutic benefit to the patients with minimal side-effects such as a feeling of paresthesia at the site of the electrodes which subsides after turning the stimulation off.

Study participants will administer non-invasive vagus nerve stimulation (nVNS) two times per day, at least five days per week, as an adjunctive therapy to their standard of care treatment for CIDP. Participants will be followed for two years to understand the impact of nVNS on CIDP symptoms and the compliance with nVNS therapies in pediatric patients.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of CIDP based upon clinical/electrophysiological criteria
* On treatment for CIDP including IVIG and/ or steroids/plasma exchange

Exclusion criteria:

* Inherited polyneuropathy, such as Charcot Tooth Marie disease
* Abnormal baseline EKG, heart disease, epilepsy, pregnancy, multiple sclerosis and diabetes mellitus

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Verma, MD, Principal Investigator — Emory University; Robert Butera, PhD, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Children's Healthcare of Atlanta, Center for Advanced Pediatrics, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta in Atlanta, Georgia, USA. Participant enrollment began February 22, 2022 and the study was terminated June 30, 2022, prior to any participant reaching the first follow-up visit at Month 6.
Groups:
- Non-invasive Vagus Nerve Stimulation (nVNS): Participants chronic inflammatory demyelinating polyneuropathy (CIDP) used the electrical neuromuscular stimulator device, VitalStim 400, while continuing to take their standard of care medication.
  Non-invasive vagus nerve stimulation (nVNS): The nVNS study intervention is delivered using a handheld electrical neuromuscular stimulator device (VitalStim 400). Participants are instructed to deliver nVNS twice per day for 60 minutes each time at least 5 days per week. The two electrodes for the device are placed on the subjects left cervical (neck) region. Parents are trained on where to place electrodes, how to ensure that the electrodes make a good contact with the skin, and how to set the stimulation parameters. The stimulation frequency (number of pulses) and amplitude (amount of current) are set during the initial baseline session in the clinic at a level that prevents discomfort and does not impact cardiorespiratory parameters. The stimulator is placed in a comfortable position, such as next to the pillow. The stimulators are battery-powered and allow configuration of the stimulation parameters to the comfort of the patient.
  Standard of care treatment: Patients are asked to continue their standard medication regimens which include in most cases will involve 3 weekly infusions of intravenous immunoglobulin (IVIG) (1 gm/kg) and rarely plasma exchange (PLEX).
Period: Overall Study
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Non-invasive Vagus Nerve Stimulation (nVNS): Participants with CIDP used the electrical neuromuscular stimulator device, VitalStim 400, while continuing to take their standard of care medication.
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Nerve Conduction Study - Distal Latency
Description: Motor nerve conduction studies are used to examine conduction of electrical impulses along nerves. Electrodes are placed on the skin in specific areas to evaluate peripheral nerves. An electrode stimulates a nerve while the receiving site records how well electrical impulses are being conducted along the nerve. Latency is the time it takes in milliseconds (ms) for the electrical impulse to travel to the site receiving the stimulation.
Time Frame: Baseline, Month 12, Month 24
Population: Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 2
ms
  Baseline | 4.8 (0.28)
  Month 12: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

2. Primary Outcome: Nerve Conduction Study - F Wave Latency
Description: Motor nerve conduction studies are used to examine conduction of electrical impulses along nerves. Electrodes are placed on the skin in specific areas to evaluate peripheral nerves. An electrode stimulates a nerve while the receiving site records how well electrical impulses are being conducted along the nerve. F wave latency is the time it takes in milliseconds (ms) for an electrical signal to travel from the stimulating electrode to the distal muscle and back to the stimulating site. F waves are used to assess polyneuropathy and F wave latency can be extended or even absent in persons with CIDP.
Time Frame: Baseline, Month 12, Month 24
Population: F wave latency was not performed for one participant at the baseline visit. Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Number; unit: ms
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 1
ms
  Baseline | 20.12
  Month 12: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

3. Primary Outcome: Nerve Conduction Study - Conduction Velocity
Description: Motor nerve conduction studies are used to examine conduction of electrical impulses along nerves. Electrodes are placed on the skin in specific areas to evaluate peripheral nerves. An electrode stimulates a nerve while the receiving site records how well electrical impulses are being conducted along the nerve. Conduction velocity measures the rate of impulse conduction in meters per second (m/s) and is often decreased in patients with CIDP as myelination is affected.
Time Frame: Baseline, Month 12, Month 24
Population: Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 2
m/s
  Baseline | 37.5 (10.61)
  Month 12: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

4. Primary Outcome: Nerve Conduction Study - Conduction Amplitude
Description: Motor nerve conduction studies are used to examine conduction of electrical impulses along nerves. Electrodes are placed on the skin in specific areas to evaluate peripheral nerves. An electrode stimulates a nerve while the receiving site records how well electrical impulses are being conducted along the nerve. Conduction amplitude is the size of the response to electrical stimulation, measured in millivolts (mV). Reduced amplitude indicates axon loss.
Time Frame: Baseline, Month 12, Month 24
Population: Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 2
mV
  Baseline | 4.15 (1.20)
  Month 12: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

5. Primary Outcome: Hand Grip Strength
Description: Hand grip strength is assessed with a Jamar Handheld Dynamometer for children ages 5-18 years and measures strength in kilograms (kg). Both right and left hand grip strength were measured and the best of three attempts were used for each hand. Increased hand strength is an indicator of effective treatment.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 2
kg
  Baseline - Right Hand | 19.1 (2.97)
  Baseline - Left Hand | 18.55 (2.62)
  Month 6 - Right Hand: number analyzed (Participants) | 0
  Month 6 - Left Hand: number analyzed (Participants) | 0
  Month 12 - Right Hand: number analyzed (Participants) | 0
  Month 12 - Left Hand: number analyzed (Participants) | 0
  Month 18 - Right Hand: number analyzed (Participants) | 0
  Month 18 - Left Hand: number analyzed (Participants) | 0
  Month 24 - Right Hand: number analyzed (Participants) | 0
  Month 24 - Left Hand: number analyzed (Participants) | 0

6. Primary Outcome: Rasch-built Overall Disability Scale (R-ODS) for CIDP Score
Description: The Rasch-built Overall Disability Scale (R-ODS) used for those with Guillain-Barré syndrome (GBS), chronic inflammatory demyelinating polyradiculoneuropathy (CIDP), and gammopathy-related polyneuropathy (MGUSP) is a 24-item scale asking respondents to rate how greatly polyneuropathy impacts activities. Responses are given on a scale of 0 to 2 where 0 indicates it is not possible for the respondent to perform the task and 2 means that the task can be performed without difficulty. Total scores range from 0 to 48 and higher scores indicate greater ability to perform daily and social tasks.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 2
score on a scale
  Baseline | 45.5 (2.12)
  Month 6: number analyzed (Participants) | 0
  Month 12: number analyzed (Participants) | 0
  Month 18: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

7. Secondary Outcome: Tumor Necrosis Factor (TNF)-α
Description: The impact of treatment on serum cytokine profiles will be assessed by measuring TNF-α. Serum cytokine levels will be statistically analyzed on a per patient basis, with each patient's baseline measurements used for comparison. TNF-α is elevated in CIDP patients and a decrease in serum TNF-α is an indication of effective treatment.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: One participant had TNF-α value at baseline that was below the limit of detection (<1.7 pg/mL) so the observation for this participant is not included as a summary score cannot be calculated. Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Number; unit: picograms per milliliter (pg/mL)
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 1
picograms per milliliter (pg/mL)
  Baseline | 2.9
  Month 6: number analyzed (Participants) | 0
  Month 12: number analyzed (Participants) | 0
  Month 18: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

8. Secondary Outcome: Interleukin (IL)-1β
Description: The impact of treatment on serum cytokine profiles will be assessed by measuring IL-1β. Serum cytokine levels will be statistically analyzed on a per patient basis, with each patient's baseline measurements used for comparison. IL-1β is elevated in CIDP patients and a decrease in IL-1β values is an indication of effective treatment.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 24
Population: One participant had a IL-1β value at baseline that was below the limit of detection (<6.5 pg/mL) so the observation for this participant is not included as a summary score cannot be calculated. Participants withdrew from the study prior to completing any follow-up study visits.
Measure: Number; unit: pg/mL
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
Number analyzed (Participants) | 1
pg/mL
  Baseline | 13.4
  Month 6: number analyzed (Participants) | 0
  Month 12: number analyzed (Participants) | 0
  Month 18: number analyzed (Participants) | 0
  Month 24: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time individuals gave consent to participate in the study until the participant withdrew from the study (up to 3 months).
Arm/Group | Non-invasive Vagus Nerve Stimulation (nVNS)
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-invasive Vagus Nerve Stimulation (nVNS) (N=2)
Tingling, numbness, and pain in limbs (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT03772717/Prot_SAP_000.pdf